CLINICAL TRIAL: NCT00575445
Title: The Use of Exhaled Nitric Oxide in Conjunction With the Asthma Control Test to Determine Asthma Control in Pediatric Patients
Status: Terminated | Type: Observational
Why Stopped: Nitric Oxide analyzer not functioning properly
Sponsor: Akron Children's Hospital (Other)
Responsible Party: Tiffany Turner, MD/Principal Investigator, Akron Children's Hospital
Other Study IDs: eNO/ACT Study
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Pediatric patients with previously diagnosed asthma

SUMMARY:
The purpose of this study is to determine if exhaled nitric oxide (eNO) levels will be increased in pediatric patients with uncontrolled asthma as determined by the Asthma Control Test (ACT). During the study the investigators will also examine if the combination of eNO and ACT will better predict asthma control that either tool alone when compared to a medical provider's assessment of the patient's asthma control.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of asthma by pediatric pulmonologist
* Age 6-18 years

Exclusion Criteria:

* Age <6 years or >18 years
* history of bronchopulmonary dysplasia
* history of cystic fibrosis
* history of primary ciliary dyskinesia
* current acute asthma exacerbation
* current acute viral upper respiratory infection
* recent ingestion of nitrate-rich foods

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric pulmonary clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Exhaled nitric oxide level | One office visit

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany L Turner, MD, Principal Investigator — Pediatric resident at Akron Children's Hospital
Locations (1):
- Akron Children's Hospital, Akron, Ohio, United States

REFERENCES:
- [Background] Meyts I, Proesmans M, De Boeck K. Exhaled nitric oxide corresponds with office evaluation of asthma control. Pediatr Pulmonol. 2003 Oct;36(4):283-9. doi: 10.1002/ppul.10317. PMID 12950039
- [Background] Nathan RA, Sorkness CA, Kosinski M, Schatz M, Li JT, Marcus P, Murray JJ, Pendergraft TB. Development of the asthma control test: a survey for assessing asthma control. J Allergy Clin Immunol. 2004 Jan;113(1):59-65. doi: 10.1016/j.jaci.2003.09.008. PMID 14713908
- [Background] Olin AC, Aldenbratt A, Ekman A, Ljungkvist G, Jungersten L, Alving K, Toren K. Increased nitric oxide in exhaled air after intake of a nitrate-rich meal. Respir Med. 2001 Feb;95(2):153-8. doi: 10.1053/rmed.2000.1010. PMID 11217912
- [Background] Malinovschi A, Janson C, Holmkvist T, Norback D, Merilainen P, Hogman M. Effect of smoking on exhaled nitric oxide and flow-independent nitric oxide exchange parameters. Eur Respir J. 2006 Aug;28(2):339-45. doi: 10.1183/09031936.06.00113705. Epub 2006 Apr 26. PMID 16641119
- [Background] Liu AH, Zeiger R, Sorkness C, Mahr T, Ostrom N, Burgess S, Rosenzweig JC, Manjunath R. Development and cross-sectional validation of the Childhood Asthma Control Test. J Allergy Clin Immunol. 2007 Apr;119(4):817-25. doi: 10.1016/j.jaci.2006.12.662. Epub 2007 Mar 13. PMID 17353040
- [Background] Lara M, Duan N, Sherbourne C, Lewis MA, Landon C, Halfon N, Brook RH. Differences between child and parent reports of symptoms among Latino children with asthma. Pediatrics. 1998 Dec;102(6):E68. doi: 10.1542/peds.102.6.e68. PMID 9832596
- [Background] Klein RB, Fritz GK, Yeung A, McQuaid EL, Mansell A. Spirometric patterns in childhood asthma: peak flow compared with other indices. Pediatr Pulmonol. 1995 Dec;20(6):372-9. doi: 10.1002/ppul.1950200607. PMID 8649917
- [Background] Hoek G, Wypij D, Brunekreef B. Self-reporting versus parental reporting of acute respiratory symptoms of children and their relation to pulmonary function and air pollution. Int J Epidemiol. 1999 Apr;28(2):293-9. doi: 10.1093/ije/28.2.293. PMID 10342694
- [Background] Grasemann H, Schwiertz R, Matthiesen S, Racke K, Ratjen F. Increased arginase activity in cystic fibrosis airways. Am J Respir Crit Care Med. 2005 Dec 15;172(12):1523-8. doi: 10.1164/rccm.200502-253OC. Epub 2005 Sep 15. PMID 16166623
- [Background] Franklin PJ, Turner SW, Mutch RC, Stick SM. Measuring exhaled nitric oxide in infants during tidal breathing: methodological issues. Pediatr Pulmonol. 2004 Jan;37(1):24-30. doi: 10.1002/ppul.10382. PMID 14679485
- [Background] Dupont LJ, Demedts MG, Verleden GM. Prospective evaluation of the validity of exhaled nitric oxide for the diagnosis of asthma. Chest. 2003 Mar;123(3):751-6. doi: 10.1378/chest.123.3.751. PMID 12628874
- [Background] Corbelli R, Bringolf-Isler B, Amacher A, Sasse B, Spycher M, Hammer J. Nasal nitric oxide measurements to screen children for primary ciliary dyskinesia. Chest. 2004 Oct;126(4):1054-9. doi: 10.1378/chest.126.4.1054. PMID 15486363
- [Background] Baraldi E, Bonetto G, Zacchello F, Filippone M. Low exhaled nitric oxide in school-age children with bronchopulmonary dysplasia and airflow limitation. Am J Respir Crit Care Med. 2005 Jan 1;171(1):68-72. doi: 10.1164/rccm.200403-298OC. Epub 2004 Oct 11. PMID 15477497
- [Background] Antus B, Csiszer E, Czebe K, Horvath I. Pulmonary infections increase exhaled nitric oxide in lung transplant recipients: a longitudinal study. Clin Transplant. 2005 Jun;19(3):377-82. doi: 10.1111/j.1399-0012.2005.00354.x. PMID 15877802